CLINICAL TRIAL: NCT02216760
Title: Determining the Pathophysiological Role of Slow Conduction Channels Identified by Ripple Mapping of the Ventricular Scar.
Brief Title: Using Ripple Mapping to Guide Substrate Ablation of Scar Related Ventricular Tachycardia.
Acronym: Ripple-VT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated prior to randomised phase
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14HH1922
Record Dates: First submitted 2014-08-07; First posted 2014-08-15 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Monomorphic Ventricular Tachycardia; Myocardial Infarction; Dilated Cardiomyopathy
Keywords: Monomorphic Ventricular Tachycardia; Myocardial infarction; Dilated cardiomyopathy; Catheter ablation; Substrate mapping; Ripple Conduction channels
MeSH Terms: conditions — Myocardial Infarction; Cardiomyopathy, Dilated

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ripple Mapping guided VT ablation (Active Comparator): Ripple Mapping (Imperial College) software (Biosense Webster) will be used to identify conduction channels within the ventricular scar substrate to guide ablation lesions in patients with monomorphic VT.
  Interventions: Device: Ripple Mapping guided VT ablation
- Conventional VT Ablation (Active Comparator): Standard substrate ablation as per local operator preference will be used to guide ablation in the ventricular scar in patients with monomorphic VT.
  Interventions: Device: Conventional VT ablation

INTERVENTIONS:
Device: Ripple Mapping guided VT ablation — RM will be used to guide identification of conduction channels and hence substrate guided ablation
  Other Names: Ripple Mapping Carto 3 V4.2 System
  Arms: Ripple Mapping guided VT ablation
Device: Conventional VT ablation — Substrate guided ablation using conventional methods (pace-mapping, LAVA/late potential abolition, scar border zone ablation)
  Arms: Conventional VT Ablation

SUMMARY:
The heart beat is controlled by electrical signals. Following a heart attack, part of the heart muscle dies and is later replaced by scar tissue. Within this area of scar, there often remain "channels" of surviving tissue still able to transmit electrical signals. However, it is well established that these "conduction channels" (CC) can form a short circuit around the scar, leading to electrical disturbances (arrhythmias) that are potentially life threatening. The commonest of these is ventricular tachycardia (VT), and is estimated to cause 300,000 deaths per year.

One recognised treatment option of VT involves burning (ablation) these "conduction channels" (CC) within the scar. However, at present, the procedure is long and is far off 100% effective. Consequently, current best practice does not rely on treating the VT, but rather preventing it from causing sudden death - this is achieved with an Implantable Cardioverter Defibrillator (ICD), a device which can recognise when a patient is in VT and deliver an internal shock to restore the normal electrical conduction. Patients with defibrillators subsequently are subject to recurrent painful and debilitating shocks which, although lifesaving, significantly reduce their quality of life. The limitation with ablation at present is due to the difficulty in visualising these CC's.

Investigators at Imperial College have created a novel electrogram visualisation program, Ripple Mapping (RM), which they have already found to be superior to currently used programmes in cases of arrhythmias in the upper chambers of the heart (the atria). During a retrospective study in patients with scar related VT following a heart attack, when ablation was delivered in areas associated with identified Ripple Mapping Conduction Channels, these patients remained free of VT recurrence for >2 year follow up interval.

The study hypothesis is that Ripple Mapping can identify all conduction channels within scar tissue critical to the VT circuit, ablation of which will lead to long-term freedom from VT and ICD therapies. The investigators now aim to perform a prospective randomised study comparing Ripple Mapping guided VT ablation against conventional VT ablation.

DETAILED DESCRIPTION:
In patients with a previous heart attack, the scar formed in the left ventricle (bottom chamber of the heart) consists of dead tissue mixed with strands of live tissue which form "conduction channels" (CC's). These Conduction channels can cause dangerous heart rhythms such as Ventricular Tachycardia (VT). This can lead to symptoms such as shortness of breath, dizziness, blackouts, and, in some, sudden death.

Patients at risk of sudden death receive special implanted devices called implantable cardioverter defibrillators (ICD) and can present with recurrent painful and debilitating ICD therapies consisting of internal shocks. Patients experiencing frequent ICD shocks due recurrent VT usually undergo a procedure to burn (ablate) the area of scar within the heart thought to be the source of the VT. This involves catheters (plastic tubes) inserted into the heart via the groin vessels allowing the cardiac electrophysiologists to obtain information about the scar. Scar tissue has low electrical voltage. By measuring the electrical voltage of the tissue in the heart, areas of scar as well as areas of live, healthy tissue can be identified and mapped. By burning (ablation) these abnormal channels of live tissue within scar (conduction channels), this can effectively reduce the episodes of VT a patient experiences, thereby reducing the frequency of shocks they experience and improve their quality of life.

In any one patient, more than 1 conduction channel and hence source of VT can be found. Current mapping technologies are incapable of providing electrophysiologists with the information that is required to locate all these conduction channels. Therefore ablation strategies have shifted from ablating in a single location in the scar, to extensive ablation within the scar in the hope that ALL conduction channels will be burnt. However, this extensive ablation strategy has no globally agreed consensus with several techniques used worldwide.

The disadvantage of this extensive ablation strategy is that the potential regions which can be responsible for VT can be large, requiring extensive ablation and therefore prolonged procedure times in sick patients who are unable to tolerate such lengthy procedures. In its current state, VT ablation by any strategy is technically challenging and time consuming with procedural times as long as 8 hours. In addition, although acute procedural success ranges from 77% to 95%, recurrence rates remain high - up to 50%.

Therefore, identification of ALL conduction channels within scar is a desirable goal for catheter ablation therapy in VT. Ripple Mapping (RM) is a novel mapping program which allows simultaneous display of "voltage" and "activation" data of the underlying ventricular tissue. RM therefore has the potential to display more detailed information of the functional properties of the underlying scar including any interspersed live tissue channels. Investigators at Imperial College have demonstrated the proof of concept of RM and validated the program in a series of abnormal heart rhythms that arise within the upper heart chambers (the atria) where RM was found to have a superior diagnostic yield as well as aiding the operator in reaching a diagnosis in shorter time when compared with conventional mapping systems. The Investigators subsequently performed a retrospective analysis of 21 patients undergoing post infarct VT ablation. All documented locations with concealed entrainment or perfect pace matches to the induced or clinical VT coincided with Ripple Mapping Conduction Channels (RMCC). In patients where ablation lesions overlapped all identified RMCCs, these patients remained free of VT recurrence for >2 year follow up interval.

The Investigators therefore propose to study the hypothesis that Ripple Mapping can identify all conduction channels within scar tissue critical to the VT circuit, ablation of which will lead to long-term freedom from VT and ICD therapies. This will be determined via a prospective randomised study comparing Ripple Mapping guided VT ablation against conventional VT ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of VT (shock/ anti tachycardia pacing/ detection) on ICD (single, dual or bi-ventricular) interrogation or 12 lead ECG.
2. Presumed scar related VT post myocardial infraction infarct/ dilated cardiomyopathy.
3. Age range 18-85yrs.
4. ICD implantation for primary or secondary prophylaxis, or device implantation pre-discharge from hospital post ablation procedure.
5. Signed informed consent

Exclusion Criteria:

1. Contraindication to catheter ablation
2. Coronary revascularisation required
3. Ventricular tachycardia due to transient, reversible causes
4. Presence of cardiac thrombus
5. Severe cerebrovascular disease
6. Active gastrointestinal disease
7. Renal failure with creatinine >200 μmol/L or on dialysis
8. Active fever or infection
9. Life expectancy shorter than the trial
10. Allergy to contrast
11. Intractable heart failure (NYHA Class IV)
12. Bleeding or clotting disorders or inability to receive heparin
13. Pregnancy
14. Must not have previous (4 weeks prior to screening) or current participation in another clinical trial with an investigational drug or investigational device
15. Unable to give informed consent
16. Unable to attend follow-up visits or ICD clinics

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Time to first appropriate ICD therapy | 24 months post ablation procedure
  There will be a 1 week post procedural blanking period. Patients will be followed up at month 3, 6, 12, 18, 24 months for ICD device interrogation post blanking interval. The presence of appropriate ICD therapy as seen on the device download will be analysed on each occasion, and the time (days) from enrollment to the study to the ICD episode will be recorded.

SECONDARY OUTCOMES:
Total appropriate ICD episodes | 24 months post ablation procedure
  There will be a 1 week post procedural blanking period. Patients will be followed up at month 3, 6, 12, 18, 24 months for ICD device interrogation post blanking interval. Appropriate ICD therapy burden (Anti-tachycardia Pacing + shocks) as well VT below the therapy zone will be recorded since the last device download and reset. The total number of episodes will be calculated and recorded for each patient at the end of 2 year follow up interval.
VT induction post procedure | 1 day
  Immediately following VT ablation, programmed ventricular stimulation will be repeated to assess whether VT is inducible. Patient outcomes will be divided into 3 groups. Group A: VT non-inducible; Group B: Non-clinical VT induced. Group C: No RMCC's identified to guide ablation OR clinical VT remains inducible. The total number of patients in each group will be calculated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Prapa Kanagaratnam, MBBChir PhD, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Hammersmith Hospital, Imperial College Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Linton NW, Koa-Wing M, Francis DP, Kojodjojo P, Lim PB, Salukhe TV, Whinnett Z, Davies DW, Peters NS, O'Neill MD, Kanagaratnam P. Cardiac ripple mapping: a novel three-dimensional visualization method for use with electroanatomic mapping of cardiac arrhythmias. Heart Rhythm. 2009 Dec;6(12):1754-62. doi: 10.1016/j.hrthm.2009.08.038. Epub 2009 Sep 3. PMID 19959125
- [Background] Jamil-Copley S, Linton N, Koa-Wing M, Kojodjojo P, Lim PB, Malcolme-Lawes L, Whinnett Z, Wright I, Davies W, Peters N, Francis DP, Kanagaratnam P. Application of ripple mapping with an electroanatomic mapping system for diagnosis of atrial tachycardias. J Cardiovasc Electrophysiol. 2013 Dec;24(12):1361-9. doi: 10.1111/jce.12259. Epub 2013 Oct 10. PMID 24118203